CLINICAL TRIAL: NCT01674244
Title: Integrative Exercise for Post-Deployment Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas C. Neylan, M.D., Professor in Residence, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-09594
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: PTSD Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrative Exercise (Experimental): Subjects will exercise for 12 weeks (3 times weekly, with each total workout being approximately 60 minutes in length). The exercise protocol will incorporate elements of mindfulness, cardiovascular strengthening, and controlled breathing.
  Interventions: Behavioral: Integrative Exercise
- Monitor Only Waitlist (Active Comparator): Monitor Only Waitlist
  Interventions: Behavioral: Monitor Only Waitlist

INTERVENTIONS:
Behavioral: Integrative Exercise
  Arms: Integrative Exercise
Behavioral: Monitor Only Waitlist
  Arms: Monitor Only Waitlist

SUMMARY:
Despite the considerable efforts of the DoD and VA to improve awareness of mental health problems and access to care, many returning veterans still report substantial barriers to seeking traditional mental health care. Research suggests that a significant barrier to pursuing treatment is the perception of stigma (Hoge at al., 2004). The primary objective of this 12-week pilot, randomized controlled trial (RCT) is to obtain pilot data on the utilization and efficacy of a standardized, integrative exercise protocol (aerobic exercise and mindful breath training) in addressing global post-traumatic stress disorder (PTSD) symptoms, sleep disturbances, and non-sleep PTSD symptoms in veterans with PTSD. Specifically, this study will examine whether a 12-week course of Integrative Exercise therapy, a treatment lacking stigma, 1) produces significant pre-post improvements in PTSD symptoms and sleep disturbances (compared to a Monitor Only Waitlist condition) 2) improves other clinical outcomes including mood, alcohol and non-alcohol substance use, psychological distress, mindfulness, and overall quality of life (compared to a Monitor Only Waitlist condition) and 3) whether such treatment is feasible and acceptable.

A secondary aim of this study is to evaluate possible mechanisms underlying these effects such as chemicals in the blood related to stress, changes in brain imaging markers, aerobic capacity, and improved sleep.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 and must be physically able to participate in an exercise program
* Participants will meet criteria for either current, full syndromal PTSD of at least 3 months duration, as indexed by the Clinician Administered PTSD Scale (CAPS) diagnostic criteria or partial PTSD defined by meeting the required number of symptoms in the B symptom cluster as well as the required number of symptoms in either the C or D symptom clusters.

Exclusion Criteria:

* Lifetime history of any psychiatric disorder with psychotic features, bipolar disorder, or mania or meet criteria for drug or alcohol dependence within the past year as assessed by the Structured Clinical Interview for DSM-IV-TR.
* Prominent suicidal or homicidal ideation
* Currently exposed to recurrent trauma or have been exposed to a traumatic event within the past 3 months
* Pregnant, have a clinically significant neurologic disorder, systemic illness affecting CNS function, history of seizure disorder, asthma, and/or physical disabilities making it impossible to use exercise equipment will be excluded
* Myocardial infarction (MI) in the past 6 months
* Moderate to severe Traumatic Brain Injury (any history of head trauma associated with the onset of persistent cognitive complaints, neurological symptoms, or loss of consciousness > 5 minutes)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) score comparison between subjects randomized to Integrative Exercise Treatment vs. Monitor Only | 12 weeks
Self-reported sleep quality comparison between subjects randomized to Integrative Exercise Treatment vs. Monitor Only | 12 weeks
Hippocampal subfield volume comparison between subjects randomized to Integrative Exercise Treatment vs. Monitor Only | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Stress and Health Research Program, University of California San Francisco, San Francisco, California, United States